CLINICAL TRIAL: NCT03395795
Title: Controlled Trial Evaluating the Interest of Noninvasive Ventilation in NAVA Mode in Respiratory Decompensations Children With Infantile Spinal Muscular Atrophy Type II
Brief Title: Trial Evaluating the Interest of Noninvasive Ventilation in NAVA Mode in Respiratory Decompensations Children With Infantile Spinal Muscular Atrophy Type II
Acronym: NAVASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160941J; IDRCB 2017-A02785-48 (Other: ANSM)
Record Dates: First submitted 2017-12-11; First posted 2018-01-10 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Infantile Spinal Muscular Atrophy
Keywords: Infantile Spinal Muscular Atrophy; Respiratory Decompensations
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Single arm trial, every patient enroll in this study will follow the same protocol with classic and NAVA mode non-invasive ventilation.
  Interventions: Device: NAVA

INTERVENTIONS:
Device: NAVA — The study has 3 phases:
  1. Phase 1:
     The patient is connected to the SERVOi® ventilator in classic VNI mode, which is parameterized according to the patient's needs and then maintained for 30min for measurements.
  2. Phase 2:
     Switch to NAVA mode (1h).
     * Definition of NAVA parameters: The positive expiratory pressure will not be modified. The NAVA level (the proportionality factor that converts the EADi (microV) to the pressure level in cmH2O was first adjusted according to the actual assisted pressure in the patient in the normal VNI mode.
     * NAVA period: The ventilatory pressure, as well as the EADI is recorded continuously for 30min after a NAVA adaptation period of about 30min.
  3. Phase 3:
  The patient returns to classic VNI mode with Phase 1 ventilatory settings for a 30 minute recording.

SUMMARY:
The new NAVA® ventilatory mode with the SERVO-i ventilator (Maquet®) uses the electrical activity of the diaphragm (EADi) as a marker for triggering the respiratory cycle. The EADi is captured by the electrodes of a specific catheter (the Edi® catheter) placed in the esophagus as a regular gastric feeding tube, and relayed to the SERVO-i who displays it and delivers respiratory assistance according to measured Edi signal which allows synchronous assistance, proportional to the respiratory efforts of the patient.

To date, no measure of the effectiveness of NAVA NAV has been performed in children with neuromuscular pathology whereas this technique could reduce the use of invasive ventilation, very iatrogenic in these fragile subjects.

DETAILED DESCRIPTION:
This is a prospective, interventional, sequential, open-label research involving ASI II children with acute respiratory decompensation requiring ventilatory support by NIV. Airway pressure, transcutaneous CO2 monitoring and hemodynamic parameters will be recorded continuously during the study, after inclusion of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age above 1 year and under 18 years
* Patient hospitalized in the pediatric intensive care unit.
* Acute respiratory decompensation requiring non-invasive ventilation for more than 6 hours.
* Patient with traditional NIV support less than 12 hours and still showing an indication for a non-invasive ventilatory support.
* Affiliation to the French health insurance organism
* Consent signed by the two holders of parental authority for the child participation in the research.

Exclusion Criteria:

* Contraindications to the use of NAVA or the setting up of a nasogastric tube.
* Hemodynamic instability requiring the use of vasopressor amines, adrenaline, norepinephrine or dobutamine.
* Severe respiratory instability requiring imminent intubation or FiO2> 60%, or PaCO2> 80 mmHg.
* Limitation of life support treatments discussed or decided.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Asynchrony percentage | At baseline
  Asynchrony percentage of non-synchronous breath cycles over all cycles of the measurement period, unaided breaths, self-initiated cycles.

SECONDARY OUTCOMES:
Feasibility | At baseline
  Frequency of obtaining an EADi signal
Feasibility | At baseline
  Percentage of effective time spent in activated NAVA mode
Efficacy and tolerance | At 30 minutes and 60 minutes
  Efficacy and tolerance: during the whole of the study period (2h30), the monitoring of transcutaneous CO2 pressure (PtcCO2) will be collected.
Efficacy and tolerance | At 30 minutes and 60 minutes
  Efficacy and tolerance: during the whole of the study period (2h30), evolution of respiratory rate will be collected.
Efficacy and tolerance | At 30 minutes and 60 minutes
  O2 saturation will be collected.
Efficacy and tolerance | At 30 minutes and 60 minutes
  FiO2 after 30 and 60 minutes under each ventilation mode will be collected.
Rate of recourse to intubation | At baseline
  Rate of recourse to intubation, patient preference.

CONTACTS AND LOCATIONS:
Overall Officials: Aben Essid, MD, Study Chair — Service de pédiatrie, Hôpital Raymond Poincaré
Locations (1):
- Service de pédiatrie, Hôpital Raymond Poincaré, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No